CLINICAL TRIAL: NCT00634998
Title: Vitamin C Supplementation as a Preventive Treatment of Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Joshua Neumiller, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10046-001; 06H-2958-9918
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Neuropathies
Keywords: Vitamin C; Ascorbic Acid; Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): 1000mg Placebo capsules orally twice daily for 90 days
  Interventions: Dietary Supplement: Placebo
- 1 (Experimental): 1000mg Vitamin C capsules orally twice daily for 90 days
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1000mg Vitamin C capsules orally twice daily
  Arms: 1
Dietary Supplement: Placebo — 1000mg Placebo capsules orally twice daily for 90 days
  Arms: 2

SUMMARY:
The purpose of this pilot study is to determine whether vitamin C supplementation is beneficial in treating and/or preventing diabetic peripheral neuropathy in people with type 2 diabetes.

DETAILED DESCRIPTION:
Painful diabetic peripheral neuropathy (DPN), a condition characterized by pain affecting the feet, legs and hands that is often characterized as burning or a "pins and needles" sensation, is estimated to affect up to 66% of the U.S. diabetic population. This pilot study will examine the effect of a daily dose of ascorbic acid, a known aldose reductase inhibitor, versus placebo, and the effect that it can have on intracellular erythrocyte (red blood cell) sorbitol levels, aldose reductase activity and aldose reductase enzyme levels utilizing benchtop methods, and effects on clinical DPN-associated pain reporting and changes in quantitative sensory testing in the lower extremities via touch discrimination and vibratory sensory testing in patients with Type 2 Diabetes Mellitus (T2DM) over the course of 90 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* diabetic peripheral neuropathy
* A1C of 6.0-10.0%

Exclusion Criteria:

* Terminal diagnosis
* Dementia
* Anemia
* Significant renal dysfunction
* History of B-12 deficiency
* Peripheral vascular disease
* Current smoker
* History of kidney stones
* Current ascorbic acid use
* Presence or foot infection and/or ulcer

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Changes in intracellular erythrocyte sorbitol levels | Changes at 90 days compared to baseline
Changes in aldose reductase enzyme activity | Activity at 90 days compared to baseline
Changes in aldose reductase enzyme levels | Levels at 90 days compared to baseline

SECONDARY OUTCOMES:
Changes in Neuropathic Pain Scale (NPS) measurement and quantitative sensory testing in the lower extremities via touch discrimination with Semmes-Weinstein monofilaments and vibratory sensation testing | Changes at 90 days compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Neumiller, PharmD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, College of Pharmacy, Department of Pharmacotherapy, Spokane, Washington, United States